CLINICAL TRIAL: NCT07162584
Title: The Modulatory Affect of Oxytocin on Human Defensive Responses During Dynamic Predator-prey Interactions
Brief Title: Oxytocin and Human Defensive Responses in a Dynamic Situation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-87
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: oxytocin; fMRI; escape decisions; dynamic predator-prey interaction; defensive responses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oxytocin group (Experimental): male and female subjects with oxytocin treatment
  Interventions: Drug: Oxytocin nasal spray
- placebo group (Placebo Comparator): male and female subjects with placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — intranasal administration of oxytocin (24 IU)
  Arms: oxytocin group
Drug: Placebo — intranasal administration of placebo (24 IU)
  Arms: placebo group

SUMMARY:
The presnet study is to investigate the effect of intranasal oxytocin (24 IU) treatment on modulating how human responsd to threat in a dynamic situation.

DETAILED DESCRIPTION:
Predator-prey interactions are inherently dynamic, requiring adaptive responses from prey to survive. Altough there is eviedence for oxytocin modulating anxiety and fear responses to threats, it remains unclear whether oxytocin (OT) would modulate how humans respond to threats along the predatory imminence continuum to facilitate escape during such interactions. Our study therefore focuses on this question by combining behavioralmeasures, skin conductance response, and fMRI in a dynamic predator-prey interaction paradigm. In this double-blind, between-subject, placebo-controlled study, participants are instructed to escape by evaluating the relative distance between themselves (i.e., the prey), the predator (slow, medium and high attacking speed) and the refuge. The MRI and Biopac electrophysiological acquisition systems are used in the study to collect subjects' brain activity and skin conductance response. Participants are also asked to rate their confidence and anxiety levels during performing the task. We will aslo examine the resulted patterns of flight initiation distance (FID) and distance to refuge (DTR) when the prey fled from different predators. Scores of questionnaires including Positive and Negative Affect Schedule, State-Trait Anxiety Inventory, Beck Depression Inventory-Ⅱ, Autism Spectrum Quotient, Sensitivity to Punishment and Sensitivity to Reward Questionnaire, General Risk Propensity Scale are also collected before the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* History of head injury; pregnant, menstruating, taking oral contraceptives; medical or psychiatric illness,
* The presence of metal in the body or claustrophobia.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Escape sucess rates when confronting different predators | 1 hour
  Escape sucess rates in successfully entering the refuge when confronting the fast, medium and slow predators.
Flight initiation distance | 1 hour
  It is the prey-predator distance when a prey flees from a threat, a key index quantifying escape decisions.
The distance to refuge | 1 hour
  The distance to refuge when a prey flees from a threat.
Brain activity patterns in response to threats along the predatory imminence continuum | 1 hour
  Brain activity patterns in response to different predators along the predatory imminence continuum. We will examine these brain response patterns via both the conventional univariate analysis and the machine learning-based multivariate pattern analysis (MVPA) approaches. Based on previous studies, the medium predator is a priori used as an anchor for fast and slow predators for a more sensitive measure of brain activity differences and contrasts with the medium predator would be reported in the suplemental files for completeness (if there were significant effects).

SECONDARY OUTCOMES:
Confidence rating scores | 1 hour
  Participants are asked to rate their confidence levels in successfully escaping from the predator before each block.
Anxiety rating scores | 1 hour
  Particioants are asked to rate how anxious they felt during the escape decision-making process.
SCR during task | 1 hour
  Skin Conductance Response (SCR) data are recorded in the task during scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Shuxia Yao, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No